CLINICAL TRIAL: NCT06507215
Title: Cross-sectional Study to Evaluate the Frequency of Dysferlinopathy Carriers in the Caucasian Population Using a Test for Detecting the Dysferlin Protein in Peripheral Blood Monocytes.
Brief Title: Dysferlinopathy Protein in Peripheral Blood Monocytes.
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MON-2011-157
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Muscular Dystrophies; Limb-Girdle Muscular Dystrophy Type 2B; Miyoshi Myopathy; Distal Myopathy With Anterior Tibial Onset
Keywords: muscular dystrophy; dysferlin; Limb-Girdle Muscular Dystrophy Type 2B; Miyoshi Myopathy; Distal Myopathy with Anterior Tibial Onset
MeSH Terms: conditions — Muscular Dystrophies; Limb-girdle muscular dystrophy, type 2B; Miyoshi myopathy; Myopathy, Distal, with Anterior Tibial Onset

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Protein analysis — The investigator enrolled 149 healthy volunteers and collected peripheral blood samples for protein analysis. While 18 of these individuals with protein levels in the range of 40%-64% were predicted to be carriers by the monocyte assay, subsequent DYSF sequencing analysis in 14 of 18 detected missense variants in only four. Analysis of DNA methylation patterns at the DYSF locus showed no changes in methylation levels at CpG islands and shores between samples.

SUMMARY:
The objective of the study is to answer the following important questions. Deficiency of the dysferlin protein is the cause of a very rare limb-girdle muscular dystrophy (LGMD-2B) that leads to significant disability. This disease is caused by mutations in the dysferlin gene. It is a recessive inherited disease, meaning that both copies of the gene must have mutations for the disease to develop. This study aims to analyze the frequency of carriers of a mutation in the DYSF gene in the Caucasian population. To achieve this, The investigator analyzed the blood of 100 healthy volunteers from their local area, quantifying the dysferlin protein in peripheral blood monocytes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with dysferlinopathies.
* Carriers of a single mutation in the DYSF gene.
* Participants who are willing to undergo treatment with oral vitamin D3.
* Subjects who can provide informed consent for participation in the study.
* Controls and carriers willing to participate in in vitro studies using HL60 cells, monocytes, and myotubes.

Exclusion Criteria:

* Individuals with conditions or medications that could interfere with the study outcomes of dysferlin expression.
* Participants who are unwilling or unable to adhere to the study protocol for the duration of the study period.
* Pregnant or breastfeeding women.
* Individuals with known allergies or adverse reactions to vitamin D3 supplements.
* Subjects with severe concurrent illnesses that may impact the study's objectives or their ability to participate effectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study focuses on individuals with dysferlinopathies, a heterogeneous group of autosomal recessive muscular dystrophies caused by mutations in the DYSF gene. It examines the effect of vitamin D3 treatment on dysferlin expression in vitro using HL60 cells, monocytes, and myotubes from controls and carriers of a single DYSF mutation. Additionally, an observational study with oral vitamin D3 in a cohort of 21 carriers demonstrates a significant increase in dysferlin expression in treated monocytes compared to untreated carriers. These findings suggest significant therapeutic implications, emphasizing the potential of combining molecular strategies with vitamin D3 supplementation to elevate dysferlin expression to non-pathological levels.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-02-27 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Dysferlin Expression Levels by age and gender | 1 month
  Dysferlin expresion lels in monocytes by western blotting

SECONDARY OUTCOMES:
Identification of Carries by Protein Level | 1 month
  Identification of Carries by Protein Level
Percentage of Predicted Carriers Showing Specific Genetic Mutations | 1 month
  Mutation Analysis of Predicted Carriers
Percentage of DNA Methylation in Target Gene | 1 month
  DNA Methylation status of the DYSF locus in order to determine wether the reduced DYSF levels in carrier and disease range had an underlying epigenetic mechanism.

CONTACTS AND LOCATIONS:
Locations (1):
- Eduard Gallardo Vigo, Barcelona, Catalonia, Spain